CLINICAL TRIAL: NCT02880618
Title: BAROSTIM THERAPY™ in Heart Failure With Reduced Ejection Fraction: A Post-Market Registry With the CE-Marked BAROSTIM NEO™ System
Brief Title: BAROSTIM THERAPY™ in Heart Failure With Reduced Ejection Fraction
Acronym: HFrEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 360049-001
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | US Export: Yes

INTERVENTIONS:
Device: Barostim Neo™ System

SUMMARY:
The purpose of this registry (NCT02880618) is to evaluate the effect of BAROSTIM THERAPY with the BAROSTIM NEO System in the commercial setting in subjects recently implanted under the CE-Marked indication for heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
Summary:

The CVRx BAROSTIM THERAPY in Heart Failure with Reduced Ejection Fraction (HFrEF) Registry will be performed with subjects who have been recently implanted with the BAROSTIM NEO System in accordance with CE-Mark approved criteria for heart failure. Subjects must be enrolled within 30 days from implant. Up to 500 subjects will be enrolled at up to 50 sites. Data should be obtained from standard of care measurements taken prior to implant, at enrollment/baseline, and at 3, 6, and 12 months after the device was implanted, at which time each subject will be exited from the registry.

Eligibility:

Subjects can be included in the Heart Failure with Reduced Ejection Fraction Registry if they were implanted in the past 30 days and meet the CE-Mark approved indications, and are not contraindicated, for the BAROSTIM NEO System in the treatment of heart failure. The BAROSTIM NEO System is indicated for subjects with heart failure, defined as New York Heart Association (NYHA) functional Class III and left ventricular ejection fraction (LVEF) ≤ 35% despite being treated with the appropriate heart failure guideline directed therapy.

The contraindications are:

* Bilateral carotid bifurcations located above the level of the mandible
* Baroreflex failure or autonomic neuropathy
* Uncontrolled, symptomatic cardiac bradyarrhythmias
* Carotid atherosclerosis that is determined by ultrasound or angiographic evaluation to be greater than 50%
* Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation

Objectives:

To describe change in the following measures at 3, 6 and 12 months compared to pre-implant baseline:

* New York Heart Association (NYHA) Class
* Six Minute Hall Walk
* Echocardiogram measures
* Biomarkers (e.g. NT-pro BNP, eGFR, Troponin HsT, Cystatin C).

Evaluate health care utilization over follow-up, such as heart failure hospitalizations.

Describe device programming and utilization

ELIGIBILITY:
Inclusion Criteria:

* Subject has heart failure, defined as New York Heart Association (NYHA) functional Class III and left ventricular ejection fraction (LVEF) ≤ 35% despite being treated with the appropriate heart failure guideline directed therapy
* Subject has been implanted with the BAROSTIM NEO System in the past 30 days
* Subject has signed an Ethics Committee approved informed consent form

Exclusion Criteria:

* Bilateral carotid bifurcations located above the level of the mandible
* Baroreflex failure or autonomic neuropathy
* Uncontrolled, symptomatic cardiac bradyarrhythmias
* Carotid atherosclerosis that is determined by ultrasound or angiographic evaluation to be greater than 50%
* Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects can be included in the Heart Failure with Reduced Ejection Fraction Registry if they were implanted in the past 30 days and meet the CE-Mark approved indications, and are not contraindicated, for the BAROSTIM NEO System in the treatment of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in New York Heart Association Functional Classification at 6 months Post-Implant | Baseline, 6 months post-implant
  To demonstrate that that treatment with BAROSTIM NEO improves New York Heart Association classification.
Change in Six Minute Hall Walk from Baseline to 6 months Post-Implant | Baseline, 6 months post-implant
  To demonstrate that that treatment with BAROSTIM NEO improves six-minute hall walk performance.
Left Ventricular Mass Index Change from Baseline to 6 Months Post-Implant | Baseline, 6 months post-implant
  To demonstrate that that treatment with BAROSTIM NEO reduces left ventricular mass index.
Change in Biomarkers from Baseline to 6 months Post-Implant (e.g. NT-pro BNP, eGFR, Troponin HsT, Cystatin C) | Baseline, 6 months post-implant
  To demonstrate that that treatment with BAROSTIM NEO improves biomarker results.
Number of Hospitalizations over Follow-Up | 12 months post-implant
  To demonstrate that that treatment with BAROSTIM NEO reduces hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Müller-Ehmsen, PhD, Study Chair — Asklepios Klinik Altona
Locations (30):
- Germany (29):
  - Herzzentrum Bad Oyenhausen, Bad Oeynhausen
  - Berlin Charité & Deutschen Herzzentrum Berlin, Berlin
  - Charité Campus Virchow Klinikum, Berlin
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Medizinisches Versorgungszentrum am Küchwald GmbH, Chemnitz
  - Universitätsklinikum Köln Herzzentrum, Cologne
  - Lippe Klinikum, Detmold
  - Dresden Friedrichstadt, Dresden
  - Herzzentrum Dresden - Interventionelle Kardiologie, Dresden
  - Herzzentrum Dresden, Elektrophysiologie, Dresden
  - Uniklinik Frankfurt, Frankfurt
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Herzzentrum Göttingen, Göttingen
  - Albertinen-Krankenhaus, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - St. Barbara Klinik Hamm, Hamm
  - Medizinische Hochschule Hannover, Hanover
  - Kardiologie im Klinikum Ingolstadt, Ingolstadt
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Herzentrum Lahr, Lahr
  - Universitätsklinikum Leipzig, Leipzig
  - Leipzig St. Georg, Leipzig
  - Universitätsklinik Mainz, Mainz
  - Clemenshospital Münster, Münster
  - St. Vincenz-Krankenhaus, Paderborn
  - Universitätsklinikum Regensburg, Regensburg
  - Marienkrankenhaus Siegen, Siegen
  - Krankenhaus & MVZ Maria-Hilf Stadtlohn GmbH, Stadtlohn
  - Klinikum Tuttlingen, Tuttlingen
- Fondazione di Ricerca e Cura "Giovanni Paolo II", Campobasso, Italy

REFERENCES:
- [Background] Abraham WT, Zile MR, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex Activation Therapy for the Treatment of Heart Failure With a Reduced Ejection Fraction. JACC Heart Fail. 2015 Jun;3(6):487-496. doi: 10.1016/j.jchf.2015.02.006. Epub 2015 May 14. PMID 25982108
- [Background] Zile MR, Abraham WT, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex activation therapy for the treatment of heart failure with a reduced ejection fraction: safety and efficacy in patients with and without cardiac resynchronization therapy. Eur J Heart Fail. 2015 Oct;17(10):1066-74. doi: 10.1002/ejhf.299. Epub 2015 Jun 10. PMID 26011593
- [Background] Gronda E, Seravalle G, Brambilla G, Costantino G, Casini A, Alsheraei A, Lovett EG, Mancia G, Grassi G. Chronic baroreflex activation effects on sympathetic nerve traffic, baroreflex function, and cardiac haemodynamics in heart failure: a proof-of-concept study. Eur J Heart Fail. 2014 Sep;16(9):977-83. doi: 10.1002/ejhf.138. Epub 2014 Jul 28. PMID 25067799
- [Background] Gronda E, Seravalle G, Trevano FQ, Costantino G, Casini A, Alsheraei A, Lovett EG, Vanoli E, Mancia G, Grassi G. Long-term chronic baroreflex activation: persistent efficacy in patients with heart failure and reduced ejection fraction. J Hypertens. 2015 Aug;33(8):1704-8. doi: 10.1097/HJH.0000000000000603. PMID 26132760
- [Background] Weaver FA, Abraham WT, Little WC, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Madershahian N, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Zile MR. Surgical Experience and Long-term Results of Baroreflex Activation Therapy for Heart Failure With Reduced Ejection Fraction. Semin Thorac Cardiovasc Surg. 2016 Summer;28(2):320-328. doi: 10.1053/j.semtcvs.2016.04.017. Epub 2016 Jun 2. PMID 28043438
- See also: BAROSTIM THERAPY — https://www.barostimtherapy.com/